CLINICAL TRIAL: NCT02727101
Title: "Rational Polytherapy" Using Perampanel Dual Therapy Anticonvulsant Combination Treatments of Adults With Refractory Focal Epilepsy : a Pilot Study.
Brief Title: Perampanel for Treatment of Adults With Refractory Focal Epilepsy : a Pilot Study.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Mid-Atlantic Epilepsy and Sleep Center, LLC (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Pavel Klein, Principle study investigator, Mid-Atlantic Epilepsy and Sleep Center, LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: maes 008
Record Dates: First submitted 2016-03-29; First posted 2016-04-04 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Epilepsy
Keywords: Focal epilepsy, Perampanel
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- phenobarbital (Active Comparator): After 12 weeks of baseline observation on phenobarbital medication, the treatment with perampanel will introduced as "add on" medication.
  Interventions: Drug: perampanel
- valproate (Active Comparator): After 12 weeks of baseline observation on valproate medication, the treatment with perampanel will introduced as "add on" medication.
  Interventions: Drug: perampanel
- lamotrigine (Active Comparator): After 12 weeks of baseline observation on lamotrigine medication, the treatment with perampanel will introduced as "add on" medication.
  Interventions: Drug: perampanel
- levetiracetam (Active Comparator): After 12 weeks of baseline observation on levetiracetam medication, the treatment with perampanel will introduced as "add on" medication.
  Interventions: Drug: perampanel
- zonisamide (Active Comparator): After 12 weeks of baseline observation on zonisamide medication, the treatment with perampanel will introduced as "add on" medication.
  Interventions: Drug: perampanel
- pregabalin (Active Comparator): After 12 weeks of baseline observation on pregabaline medication, the treatment with perampanel will introduced as "add on" medication.
  Interventions: Drug: perampanel
- lacosamide (Active Comparator): After 12 weeks of baseline observation on lacosasmide medication, the treatment with perampanel will introduced as "add on" medication.
  Interventions: Drug: perampanel
- clobazam (Active Comparator): After 12 weeks of baseline observation on clobazam medication, the treatment with perampanel will introduced as "add on" medication.
  Interventions: Drug: perampanel
- ezogabine (Active Comparator): After 12 weeks of baseline observation on ezogabine medication, the treatment with perampanel will introduced as "add on" medication.
  Interventions: Drug: perampanel
- eslicarbazepine (Active Comparator): After 12 weeks of baseline observation on eslicarbamazepine medication, the treatment with perampanel will introduced as "add on" medication.
  Interventions: Drug: perampanel
- topiramate (Active Comparator): After 12 weeks of baseline observation on eslicarbamazepine medication, the treatment with perampanel will introduced as "add on" medication.
  Interventions: Drug: perampanel
- tiagabine (Active Comparator): After 12 weeks of baseline observation on eslicarbamazepine medication, the treatment with perampanel will introduced as "add on" medication.
  Interventions: Drug: perampanel

INTERVENTIONS:
Drug: perampanel — Each group of 6 patients will be followed for 12 weeks of baseline observation on baseline medication. Seizure frequency will be counted, using subjects' self-reported seizure diaries. Perampanel will be titrated to 8-12 mg/day, with the final dose determined by side effects and tolerability of Perampanel at 8-12 mg/day doses. Titration will occur at the rate of 2 mg/week or two weeks, as tolerated.
  Other Names: Fycompa

SUMMARY:
The goal of the present study is to evaluate ("screen") a large number (12) of different dual therapies of perampanel + another AED ("PMP+") for a large, 75-100% seizure frequency reduction. The design of the study will differ from usual AED studies. The study will be (i) open label, with (ii) a small n per group, n=6, with (iii) outcome measures a 'blockbuster effect': (a) ≥75 seizure frequency reduction; and (b) seizure freedom.

DETAILED DESCRIPTION:
Investigators will compare rates of seizure freedom and >75% seizure frequency reduction among 12 treatment arms consisting of 6 subjects each with refractory focal epilepsy treated with perampanel and one other AED ("PMP+"). Treatment arms will include (1) Perampanel +phenobarbital, (2) PMP+valproate, (3) PMP+ lamotrigine, (4) PMP + topiramate, (5) PMP + tiagabine, (6) PMP + levetiracetam, (7) PMP + zonisamide, (8) PMP + pregabalin, (9) PMP + lacosamide, (10) PMP+ clobazam, (11) PMP + ezogabine; and (12) PMP + eslicarbazepine. Each group of 6 will be followed for 12 weeks of baseline observation on baseline medication. Seizure frequency will be counted, using subjects' self-reported seizure diaries. PMP will be titrated to 8-12 mg/day, with the final dose determined by side effects and tolerability of PMP at 8-12 mg/day doses. Titration will occur at the rate of 2 mg/week or two weeks (in accordance with FDA labeling), as tolerated. Subjects will be observed for 12 weeks of maintenance treatment on the target PMP doses. Seizure frequency will be compared between the 12 weeks of baseline observation and 12 weeks of maintenance treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Stable focal epilepsy, with partial complex seizures including partial complex seizures with or without secondary generalization, partial simple seizures with a clear motor component with or without secondary generalization, and partial simple seizures with secondary generalization.
3. Stable dose for at least 30 days of the chosen background AED dose
4. Epilepsy duration for > 2 years
5. Past/current treatment with > 4 AEDs. Vagal nerve stimulator treatment will be allowed and will not count as an AED. VNS setting must be stable for 3 months prior to enrollment.
6. Seizure frequency of ≥1/month

Exclusion Criteria:

1. Primary generalized epilepsy
2. Simple partial seizures without motor components or secondary generalization
3. Non-epileptic seizures
4. Progressive neurological disease including growing neoplasm, CNS degenerative disorders including Alzheimer's disease, other forms of dementia
5. Any systemic illness or unstable medical condition that might pose additional risk, including renal or liver disease, clinically uncontrolled cardiac disease, other unstable metabolic or endocrine disturbances, and active systemic cancer
6. Change in the dose of any Antiepileptic Drug within 30 days prior to enrollment
7. Psychosis within six months of enrollment.
8. Active drug or alcohol dependence or any other factors that, in the opinion of the site investigators would interfere with adherence to study requirements;
9. Pregnancy
10. Use of any CNS-active investigational drugs within 3 months of enrollment.
11. Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-11; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
responder rate | 12 weeks
  responder rate, defined by >75% seizure frequency reduction. Average seizure frequency per 4 weeks will be compared between the 12 weeks of "PMP+" maintenance treatment and 12 weeks of baseline.
seizure freedom rate | 12 weeks
  seizure freedom rate. Proportion of responders and of subjects with seizure freedom in each treatment arm will be compared with historical data of 75% seizure reduction from pivotal phase 3 studies for which such data is publicly available
treatment discontinuation rate | 12 weeks
  To evaluate the safety and tolerability of each perampanel+ combination with treatment discontinuation rate as the primary safety/tolerability outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Klein, M.B,B.Chir., Principal Investigator — Mid-Atlantic Epilepsy and Sleep Center
Locations (1):
- MidAtlantic Epilepsy and Sleep Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided